CLINICAL TRIAL: NCT02363673
Title: The Effect of Individualised Homoeopathic Treatment of Autism Spectrum Disorder in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Johannesburg (Other)
Responsible Party: Principal Investigator, Dr J. Pellow, Dr J. Pellow, University of Johannesburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGoodwin201006636; REC-01-128-2014 (Other: University of Johannesburg)
Record Dates: First submitted 2015-02-09; First posted 2015-02-16 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Children; Homoeopathy
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Individualised Homoeopathic Remedy (Experimental): Each participant is to receive an individualised homoeopathic remedy in aqua distilla according to their symptoms and characteristic manifestations of their disorder. Although different individualised remedies may be dispensed, each remedy will be homoeopathic. Remedies will be dispensed in aqua distilla. Each individualised homoeopathic remedy will have an individualised dosage, frequency and duration based on the laws of individualised homoeopathic prescribing.
  Interventions: Other: Individualised homoeopathic remedy in aqua distilla

INTERVENTIONS:
Other: Individualised homoeopathic remedy in aqua distilla — Each participant is to receive an individualised homoeopathic remedy according to their symptoms and characteristic manifestations of their disorder.

SUMMARY:
The aim of this study is to determine the effect of individualised homoeopathic treatment of children with Autism Spectrum Disorder (ASD).This study is of descriptive case study design, with a structured interview and quantitative measurement components taking place over 12 weeks, with a consultation every 4 weeks. Children aged 3-6 years of age with ASD are invited to participate and their parent/guardian is required to be present during each consultation. Each consultation will consist of a homoeopathic case taking, conduction of the Childhood Autism Rating Scale (CARS) and Autism Treatment Evaluation Checklist (ATEC) measures and a brief physical exam. After each consultation, the participant will receive an individualised homoeopathic remedy, according to their individual symptoms and characteristics, to take for the subsequent 4 weeks. This remedy will be determined using the Mercurius® repertory software.

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of individualised homoeopathic treatment of children with Autism Spectrum Disorder (ASD). A minimum of 10 participants between the ages of 3 to 6 years, both male and female, will be recruited. This study is of a descriptive case study design, with a structured interview and quantitative measurement components. The data collection will take place over 12 weeks at both the University of Johannesburg's Health Training Centre and the schools for Autistic children within Gauteng.

A parent/guardian must be present for all consultations to aid data collection. Week 0 will consist of an explanation of the study, the Participant Information and Assent Form and the Parent/Guardian Information Form . The Consent Form will be signed by the parent or guardian if they wish their child to participate in the study. The child will also be informed on the details of the study and have to consent to their participation.

The participant will be screened using screening checklist, which includes the completion of the CARS by the researcher and guardian, to determine their eligibility to take part in the research study. If they are eligible to take part in the study, the researcher will conduct a case taking, the ATEC and a relevant physical examination (including vital signs). This information will serve as a baseline for each participant in the study along with the previous information attained from the CARS used in the participant's screening.

The first interview will consist of a structured interview of approximately 90 minutes duration with the parent/guardian, where after the following structured interviews will take 60 minutes, wherein the participant will be free to move around and interact with their environment as naturally as possible.

The researcher will then establish the participant's individualised homoeopathic remedy according to the principles of classical homoeopathy by using the Complete Repertory 2014 provided in Mercurius® repertory software.The selected remedy will be provided to the participant within 24 hours with instruction on how to take it.

The participant will be consulted with their parent/guardian 3 more times, at weeks 4, 8 and 12, where on each occasion they will have their case taken, the CARS and the ATEC conducted as well as a relevant physical examination. At the interviews on week 4 and 8, each case will be re-evaluated and the appropriate individualised homoeopathic remedy dispensed. Each participant will receive their individualised homoeopathic remedy in aqua distilla drops to be put into the participant's mouth, which will be prescribed with the most suitable repetition and potency for the participant, according to laws of homoeopathy that govern individualised homoeopathic prescribing. The case taking will assist in determining the potency and frequency of the remedy given. No remedy will be dispensed at week 12.

Data will be analysed by Statkon using non-parametric tests including the Friedman and the Wilcoxin post-hoc analyses. A positive outcome of this study will contribute to the accessibility of a complementary treatment for ASD as well as denote the requirement for further research studies on the subject. The outcome of this study may add to the body of knowledge of individualised homoeopathic treatment on ASD.

ELIGIBILITY:
Inclusion Criteria:

* children aged of 3 to 6 years;
* diagnosed with ASD by a physician, psychologist, psychiatrist or neurologist;
* are on no medication or are on medication for ASD and its comorbid conditions for more than 2 months;
* are able to have their guardian present for all interviews, and
* have mild-to-moderate symptoms ASD as measured using the CARS

Exclusion Criteria:

* a history of or contract organic brain damage, meningitis, epilepsy or encephalitis;
* are on conventional medication such as Fluoxetine, Methylphenidate, Atomoxetine or Risperidal for less than 2 months or make use of any new medication for ASD or its comorbid conditions for the duration of the study, or
* currently be taking any herbal or homoeopathic medications.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale | Every 4 weeks for 12 weeks
  The Childhood Autism Rating Scale will be conducted at weeks 0, 4, 8 and 12.

SECONDARY OUTCOMES:
Autism Treatment Evaluation Checklist | Every 4 weeks for 12 weeks
  The Autism Treatment Evaluation Checklist will be conducted at weeks 0, 4, 8 and 12.
Case notes | Every 4 weeks for 12 weeks
  Qualitative data collection will be collect by means of case notes which will be taken at weeks 0, 4, 8 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: N Gower, MTechHom, Study Director — Senior Lecturer
Locations (1):
- University of Johannesburg Doornfontein Campus, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No